CLINICAL TRIAL: NCT03750786
Title: A Randomized, Multicenter, Parallel-group, Phase III Study to Compare the Efficacy of Arfolitixorin Versus Leucovorin in Combination With 5 Fluorouracil, Oxaliplatin, and Bevacizumab in Patients With Advanced Colorectal Cancer
Brief Title: A Study to Compare the Efficacy of Arfolitixorin Versus Leucovorin in Combination With 5 Fluorouracil, Oxaliplatin, and Bevacizumab in Patients With Advanced Colorectal Cancer
Acronym: AGENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isofol Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISO-CC-007
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Leucovorin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): ARFOX (Arfolitixorin and 5-FU and Oxaliplatin) and Bevacizumab
  Interventions: Drug: Arfolitixorin
- Group B (Active Comparator): mFOLFOX-6 (Leucovorin and 5-FU and Oxaliplatin) and Bevacizumab
  Interventions: Drug: Leucovorin

INTERVENTIONS:
Drug: Arfolitixorin — Bevacizumab 5 mg/kg intravenous infusion; Oxaliplatin 85 mg/m2 intravenous infusion; 5-FU 400 mg/m2 intravenous bolus; Arfolitixorin 60 mg/m2 intravenous bolus; 5-FU 2400 mg/m2 intravenous infusion; Arfolitixorin 60 mg/m2 intravenous bolus
  Arms: Group A
Drug: Leucovorin — Bevacizumab 5 mg/kg intravenous infusion; Oxaliplatin 85 mg/m2 intravenous infusion; Leucovorin 400 mg/m2 intravenous infusion; 5-FU 400 mg/m2 intravenous infusion; 5-FU 2400 mg/m2 intravenous infusion
  Arms: Group B

SUMMARY:
This is a multicenter, randomized, parallel-group, Phase III study in at least 440 patients with advanced colorectal cancer to compare the efficacy of treatment with arfolitixorin versus Leucovorin in combination with 5-fluorouracil, oxaliplatin, and bevacizumab according to modified FOLFOX-6 until PD according to RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal adenocarcinoma verified by biopsy.
2. Availability of biopsy material, from the primary tumor or metastasis, allowing for analysis of tumor gene expression.
3. Non-resectable metastatic CRC planned for first line therapy with 5-FU, Leucovorin, oxaliplatin, and bevacizumab.
4. Evaluable disease with at least one measurable lesion of metastatic disease (≥10 mm in longest diameter on axial image on CT-scan or alternatively MRI with <5 mm reconstruction interval) or lymph node (≥ 15 mm in shortest axis when assessed by CT) obtained within 28 days of randomization.
5. Life expectancy of more than 4 months.
6. ECOG performance status 0 or 1.
7. Hemoglobin (Hb) > 80 g/L, Absolute neutrophil count (ANC) > 1.5x10E9/L. Thrombocytes > 100x10E9/L.
8. Creatinine clearance > 50 mL/min, Total bilirubin < 1.5 x ULN, AST and ALT < 3 x ULN (and < 5 x ULN in case of liver metastases).
9. Male or female ≥18 years of age.
10. Female patients of childbearing potential must have a negative urine pregnancy test and use adequate contraceptive measures . Male patients must use adequate contraceptive measures .
11. Voluntarily signed informed consent before performance of any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Malignant tumors other than colorectal adenocarcinomas (current or within the previous five years), with the exception for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix.
2. Less than 6 months between randomization and completion of the last anti-cancer treatment (chemotherapy/radiotherapy/immunotherapy, etc.). (NB: Rectal cancer treatment shorter than 8 weeks of chemo/radiation therapy is allowed.)
3. Confirmation of progressive disease within 6 months after completion of prior adjuvant anti-cancer treatment.
4. Indication for any metastatic Colo-rectal Cancer (mCRC) surgery or anti-cancer treatment other than study treatment.
5. Prior treatment with arfolitixorin.
6. Indication for treatment with a 5-FU analogue, or 5-FU for a condition other than mCRC.
7. Known Dihydropyrimidine Dehydrogenase Deficiency (DPD) deficiency.
8. Known or suspected central nervous system (CNS) metastases.
9. Unresolved bowel obstruction, uncontrolled Crohn's disease, or ulcerative colitis.
10. History of cardiac disease with a New York Heart Association Class II or greater, congestive heart failure, myocardial infarction, or unstable angina at any time during the 6 months prior to randomization, or serious arrhythmias requiring medication for treatment.
11. Current CTCAE ≥ grade 3 diarrhea.
12. Current chronic infection or uncontrolled serious illness causing immunodeficiency.
13. Known or suspected hypersensitivity or intolerance to arfolitixorin, LV, 5-FU, oxaliplatin, or bevacizumab.
14. Breastfeeding patients.
15. Patient who received investigational drugs in other clinical trials within 28 days, or 5 half-lives of the investigational drug, prior to randomization.
16. Patient with serious medical or psychiatric illness likely to interfere with participation in this clinical study.
17. Ongoing drug or alcohol abuse, as deemed by the Investigator.
18. Any condition that, in the opinion of the Investigator, could compromise the patient's safety or adherence to the study protocol.
19. Involvement, or related to people involved in the planning or conduct of the study (applies to both Isofol Medical AB (publ) staff and staff at the study site)
20. Surgery (excluding previous diagnostic biopsy) in the 28-day period before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, Prof., Principal Investigator — Vall d'Hebron Institute of Oncology
Locations (94):
- United States (18):
  - 840-24 - Banner Gateway Medical Center, Gilbert, Arizona
  - 840-15 - University of Southern California, Los Angeles, California
  - 840-01 - HOAG Memorial Hospital, Newport Beach, California
  - 840-13 - UCH-MHS d/b/a Memorial Health System, Colorado Springs, Colorado
  - 840-34 - Banner MD Anderson Cancer Center, Greeley, Colorado
  - 840-32 - University of Miami, Miami, Florida
  - 840-08 - Pinellas Hematology Oncology, St. Petersburg, Florida
  - 840-30 - Joliet Oncology-Hematology Associates, Joliet, Illinois
  - 840-06 - Cancer Center of Kansas, Wichita, Kansas
  - 840-29 - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - 840-19 - University of Louisville Research Foundation Inc. (ULRF), Louisville, Kentucky
  - 840-14 - University of Michigan Cancer Center, Ann Arbor, Michigan
  - 840-04 - St. Vincent Frontier Cancer Center, Billings, Montana
  - 840-12 - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - 840-22 - University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma
  - 840-10 - Oregon Health and Science University-Knight Cancer Institute, Portland, Oregon
  - 840-27 - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - 840-02 - The University of Texas Health Science Center, San Antonio, Texas
- Australia (8):
  - 036-10 - Border Medical Oncology Research Unit, Albury, New South Wales
  - 036-02 - Chris O'Brien Lifehouse, Sydney, New South Wales
  - 036-03 - Westmead Hospital, Sydney, New South Wales
  - 036-09 - Southern Medical Day Care Center, Wollongong, New South Wales
  - 036-04 - Peninsula Health - Frankston Hospital, Frankston, Victoria
  - 036-01 - Western Health - Sunshine Hospital, Melbourne, Victoria
  - 036-07 - Northern Health - Epping Hospital, Melbourne, Victoria
  - 036-05 - Monash Health, Melbourne, Victoria
- Austria (6):
  - 040-02 - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - 040-06 - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
  - 040-03 - Uniklinikum Salzburg, Salzburg
  - 040-01 - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - 040-05 - Wilhelminenspital, Vienna
  - 040-04 - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Canada (10):
  - 124-03 - William Osler Health System - Brampton Civi Hospital, Brampton, Ontario
  - 124-10 - Thunder Bay Regional Health Research Institute, Thunder Bay, Ontario
  - 124-07 - Sunnybrook Research Institute, Toronto, Ontario
  - 124-04 - CISSS de l'Outaouais - Hôpital de Gatineau, Gatineau, Quebec
  - 124-11 - CISSS de Chaudière-Appalaches, Lévis, Quebec
  - 124-01 - Montreal University Health Center, Montreal, Quebec
  - 124-02 - Hôpital de la Cité-de-la-Santé, Laval
  - 124-08 - Hôpital Maisonneuve Rosemont, Montreal
  - 124-06 - Jewish General Hospital, Montreal
  - 124-05 - Ottawa Hospital Research Institute, Ottawa
- France (9):
  - 250-07 - Hôpital Henri Mondor, Créteil
  - 250-06 - Centre Georges Francois Leclerc, Dijon
  - 250-01 - Institute Hospitalier Franco-Britannique, Levallois-Perret
  - 250-09 - Hopital Privé Jean Mermoz, Lyon
  - 250-08 - Hôpital Européen, Marseille
  - 250-03 - Hôpital Paris Saint Joseph, Paris
  - 250-02 - Hôpital Saint-Antoine, Paris
  - 250-04 - Polyclinique Francheville, Périgueux
  - 250-05 - Clinique Sainte Anne, Strasbourg
- Germany (12):
  - 276-12 - Charité - Universitätsmedizin Berlin, Berlin
  - 276-02 - Universitätsklinikum Carl Gustav Carus, Dresden
  - 276-03 - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - 276-10 - Universitärers Cancer Center Hamburg (UCCH), Hamburg
  - 276-11 - Klinikum Kassel GmbH, Kassel
  - 276-04 - MVZ Mitte - Onkologische Schwerpunktpraxis, Leipzig
  - 276-13 - Universitäres Krebszentrum Leipzig (UCCL), Leipzig
  - 276-07 - Philipps-Universität Marburg, Marburg
  - 276-08 - Carl von Basedow Klinikum Saalekrei GmbH, Merseburg
  - 276-01 - Klinikum der Universität München - Campus Grosshadern, München
  - 276-09 - Klinikum Nürnberg Nord, Nuremberg
  - 276-05 - Kliniken Nordoberpfalz AG, Weiden
- Greece (6):
  - 300-04 - 251 Airforce Hospital, Athens
  - 300-01 - Aretaieo Hospital, Athens
  - 300-02 - University General Hospital Attikon, Athens
  - 300-03 - Metropolitan General Hospital, Athens
  - 300-05 - Metropolitan General SA, Athens
  - 300-06 - University General Hospital of Larissa, Larissa
- Japan (15):
  - 392-10 - Aichi Cancer Center, Aichi
  - 392-01 - National Cancer Center Hospital East, Chiba
  - 392-09 - National Hospital Organization Shikoku Cancer Center, Ehime
  - 392-07 - Gifu University Hospital, Gifu
  - 392-12 - Saitama Medical University International Medical Center, Hidaka
  - 392-05 - University of Tsukuba Hospital, Ibaraki
  - 392-15 - Kagawa University Hospital, Kagawa
  - 392-08 - St.Marianna University School of Medicine Hospital, Kanagawa
  - 392-11 - National Hospital Organization Osaka National Hospital, Osaka
  - 392-13 - Osaka General Medical Center, Osaka
  - 392-14 - Kansai Medical University Hospital, Osaka
  - 392-04 - Saitama Cancer Center, Saitama
  - 392-03 - Hokkaido University Hospital, Sapporo Hokkaido
  - 392-02 - Shizuoka Cancer Center, Shizuoka
  - 392-06 - National Cancer Center Hospital, Tokyo
- Spain (8):
  - 724-03 - Instituto Oncologico Baselga - Hospital Quiron, Barcelona
  - 724-07 - Hospital del la Santa Creu i Sant Pau, Barcelona
  - 724-01 - Vall d'Hebron Institute of Oncology, Barcelona
  - 724-06 - Hospital Universitario Reina Sofia, Córdoba
  - 724-04 - Hospital Unviersitario 12 de Octubre, Madrid
  - 724-09 - Hospital Universitario HM Sanchinarro, Madrid
  - 724-02 - Hospital Regional Universitario Carlos Haya, Málaga
  - 724-05 - Hospital Universitario Virgen del Rocío, Seville
- Sweden (2):
  - 752-02 - Södersjukhuset, Stockholm
  - 752-01 - Akademiska Sjukhuset, Uppsala

REFERENCES:
- [Derived] Tabernero J, Yoshino T, Stintzing S, de Gramont A, Gibbs P, Jonker DJ, Nygren P, Papadimitriou C, Prager GW, Tell R, Lenz HJ. A Randomized Phase III Study of Arfolitixorin versus Leucovorin with 5-Fluorouracil, Oxaliplatin, and Bevacizumab for First-Line Treatment of Metastatic Colorectal Cancer: The AGENT Trial. Cancer Res Commun. 2024 Jan 4;4(1):28-37. doi: 10.1158/2767-9764.CRC-23-0361. PMID 38059497

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: ARFOX (Arfolitixorin and 5-FU and Oxaliplatin) and Bevacizumab
  Arfolitixorin: Arfolitixorin and 5-FU and Oxaliplatin and Bevacizumab
- Group B: mFOLFOX-6 (Leucovorin and 5-FU and Oxaliplatin) and Bevacizumab
  Leucovorin: Leucovorin and 5-FU and Oxaliplatin and Bevacizumab
Period: Overall Study
Arm/Group | Group A | Group B
Started | 245 | 245
Completed | 0 | 0
Not Completed | 245 | 245

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 245 | 245 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (10.5) | 62.6 (10.7) | 62.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 94 | 177
  Male | 162 | 151 | 313
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 204 | 214 | 418
  Unknown or Not Reported | 41 | 31 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 36 | 35 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 179 | 192 | 371
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 30 | 18 | 48
Time since initial diagnosis, months [Mean (Standard Deviation); unit: months] | 9.7 (20.9) | 7.7 (15.2) | 8.7 (18.1)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Best ORR, defined as the best response recorded from the start of the study treatment until the end of treatment.
Time Frame: Until disease progression, an average of ten months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 245 | 245
Participants
  Complete Response | 2 | 5
  Partial Response | 116 | 116
  Stable Disease | 106 | 86
  Progressive Disease | 7 | 11
  Non-CR/Non-PD | 6 | 3
  No BOR Available | 6 | 18
  Not Evaluable | 2 | 6

2. Secondary Outcome: Progression Free Survival
Description: PFS, defined as the time from randomization to first occurrence of tumor progression based on CT-scans/MRIs.
Time Frame: Until disease progression, an average of ten months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A | Group B
Number analyzed (Participants) | 245 | 245
months | 12.8 [10.9 to 13.2] | 11.6 [11.0 to 14.5]

3. Secondary Outcome: Duration of Response
Description: The duration of response is measured from the time measurement criteria are first met for CR/PR until the first date that recurrent or progressive disease is objectively documented.
Time Frame: Until disease progression, an average of ten months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A | Group B
Number analyzed (Participants) | 118 | 121
months | 12.2 [11.1 to 14.1] | 12.9 [10.6 to 15.0]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 118/243 | 100/238
Serious Adverse Events (participants affected / at risk) | 81/243 | 86/238
Other Adverse Events (participants affected / at risk) | 239/243 | 231/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=243) | Group B (N=238)
Enterococcal Infection (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1
Escherichia Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Intestinal Fistula Infection (Infections and infestations) | 1 | 0
Klebsiella Infection (Infections and infestations) | 1 | 0
Liver Abscess (Infections and infestations) | 0 | 1
Pelvic Abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia Viral (Infections and infestations) | 1 | 0
Pulmonary Sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 3
General Physical Health Deterioration (General disorders) | 1 | 3
Catheter Site Extravasation (General disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Condition Aggravated (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 5
Anemia (Blood and lymphatic system disorders) | 2 | 1
Hemolytic Anemia (Blood and lymphatic system disorders) | 1 | 0
Leukaemoid Reaction (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0
Stoma Site Hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 3
Urinary Retention (Renal and urinary disorders) | 1 | 2
Renal Colic (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Atrial Thrombosis (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Low Cardiac Output Syndrome (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Acidosis Hyperchloremic (Metabolism and nutrition disorders) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Lactic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Metabolic Encephalopathy (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Peroneal Nerve Palsy (Nervous system disorders) | 1 | 0
Status Epilepticus (Nervous system disorders) | 1 | 0
Transient Ischemic Attack (Nervous system disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 2
Biliary Fistula (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Portosplenomesenteric Venous Thrombosis (Hepatobiliary disorders) | 0 | 1
Depp Vein Thrombosis (Vascular disorders) | 2 | 0
Embolism Arterial (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Superior Vena Cava Syndrome (Vascular disorders) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
C-Reactive Protein Increased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertrophic Cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 1
Anaphylactic Shock (Immune system disorders) | 0 | 1
Rectoprostatic Fistula (Reproductive system and breast disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 2 | 1
Crohn's Disease (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 6 | 10
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Intra-Abdominal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 5 | 4
Large Intestine Perforation (Gastrointestinal disorders) | 3 | 2
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Melena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 2
Rectal Perforation (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 5
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0
Abdominal Sepsis (Infections and infestations) | 1 | 0
Abdominal Wall Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacteremia (Infections and infestations) | 0 | 1
Biliary Tract Infection (Infections and infestations) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 1 | 0
Corona Virus Infection (Infections and infestations) | 3 | 1
Ecthyma (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 3 | 3
Septic Shock (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 4
Urosepsis (Infections and infestations) | 0 | 2
Device Related Infection (Infections and infestations) | 3 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=243) | Group B (N=238)
Neurotoxicity (Nervous system disorders) | 40 | 22
Dizziness (Nervous system disorders) | 23 | 20
Polyneuropathy (Nervous system disorders) | 16 | 16
Hypoaesthesia (Nervous system disorders) | 11 | 18
Dyspepsia (Gastrointestinal disorders) | 12 | 23
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 20 | 12
Abdominal Pain Upper (Gastrointestinal disorders) | 16 | 14
Malaise (General disorders) | 13 | 13
Oedema Peripheral (General disorders) | 13 | 8
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 21 | 19
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Weight Decreased (Investigations) | 22 | 20
Aspartate Aminotransferase Increased (Investigations) | 22 | 13
Alanine Aminotransferase Increased (Investigations) | 23 | 11
Gamma-glutamyltransferase Increased (Investigations) | 14 | 17
Blood Alkaline Phosphatase Increased (Investigations) | 9 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 28
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 16
Dry Skin (Skin and subcutaneous tissue disorders) | 13 | 21
Rash (Skin and subcutaneous tissue disorders) | 12 | 13
Back Pain (Musculoskeletal and connective tissue disorders) | 23 | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 11
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 11 | 13
Proteinuria (Renal and urinary disorders) | 23 | 13
Insomnia (Psychiatric disorders) | 11 | 18
Depression (Psychiatric disorders) | 5 | 13
Anemia (Blood and lymphatic system disorders) | 44 | 51
Neutropenia (Blood and lymphatic system disorders) | 60 | 51
Thrombocytopenia (Blood and lymphatic system disorders) | 32 | 28
Abdominal Pain (Gastrointestinal disorders) | 51 | 50
Constipation (Gastrointestinal disorders) | 69 | 64
Diarrhea (Gastrointestinal disorders) | 118 | 113
Nausea (Gastrointestinal disorders) | 117 | 123
Stomatitis (Gastrointestinal disorders) | 52 | 62
Vomiting (Gastrointestinal disorders) | 60 | 55
Asthenia (General disorders) | 48 | 42
Fatigue (General disorders) | 108 | 103
Mucosal Inflammation (General disorders) | 53 | 49
Pyrexia (General disorders) | 45 | 39
Urinary Tract Infection (Infections and infestations) | 24 | 27
Neutrophil Count Decreased (Investigations) | 53 | 62
Platelet Count Decreased (Investigations) | 33 | 35
White Blood Cell Count Decreased (Investigations) | 24 | 25
Decreased Appetite (Metabolism and nutrition disorders) | 66 | 60
Dysesthesia (Nervous system disorders) | 26 | 31
Dysgeusia (Nervous system disorders) | 40 | 37
Headache (Nervous system disorders) | 25 | 24
Neuropathy Peripheral (Nervous system disorders) | 73 | 64
Paresthesia (Nervous system disorders) | 36 | 42
Peripheral Sensory Neuropathy (Nervous system disorders) | 66 | 72
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 64 | 62
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 32
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 20 | 29
Hypertension (Vascular disorders) | 55 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT03750786/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT03750786/SAP_001.pdf